CLINICAL TRIAL: NCT00976079
Title: The Effect of Transcutaneous Electrical Nerve Stimulation on Quadriceps Central Activation and Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Christopher D. Ingersoll, PhD, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13360
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2009-09-14 (Estimated); Status verified 2009-09

CONDITIONS: Tibial Femoral Knee Osteoarthritis; Osteoarthritis
Keywords: Tibial femoral knee osteoarthritis; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active TENS (Experimental): Active TENS therapy for 4 weeks plus standard physical therapy for same time period.
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)
- Placebo TENS (Placebo Comparator): Placebo TENS for 4 weeks plus standard physical therapy for same time period.
  Interventions: Device: Placebo TENS
- Control Group (No Intervention): No TENS, standard physical therapy for 4 weeks.

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — Continuous TENS use
  Arms: Active TENS
Device: Placebo TENS — Placebo TENS use
  Arms: Placebo TENS

SUMMARY:
Participants diagnosed with tibial femoral knee osteoarthritis will be assigned to one of three treatment groups including: active transcutaneous electrical nerve stimulation (TENS), placebo TENS, and a control group. Assignment of conditions will be concealed. All participants in each of the three groups will receive physical therapy for all 4 weeks of the intervention. Main outcome measures will include quadriceps central activation ratio, quadriceps torque production, WOMAC scores, visual analog pain scores during gait as well as knee joint kinetics and kinematics during gait. The purpose of this study is to to determine if the continuous use of TENS therapy for activities of daily living and rehabilitation will positively impact all outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with a Kellgren and Lawrence grade of 1- 4 for Tibial Femoral Knee OA in at least one leg or have been diagnosed with OA by a physician using evidence confirmed from imaging studies, arthroscopy, or visualization during an past surgical procedures, or have medical reports confirming OA using imaging studies, arthroscopy, or visualization during an past surgical procedures.
* Patients between the ages of 18 and 80 years of age.
* Patients will have a CAR less than 90%.

Exclusion Criteria:

* Patients who are pregnant.
* Patients who have sought medical attention for a trauma to the knee injury within the past 6 months.
* Patients who have had any orthopaedic lower extremity surgery in the past 6 months, or any surgery that would inhibition proper functioning of the study methodology.
* Patients with a diagnosis of Rheumatoid Arthritis.
* Patients with a known hypersensitivity to electrical stimulation.
* Patients with any types of neuropathy.
* Patients with known muscular abnormalities.
* Patients with a history of a heart condition that precludes them from exercise.
* The technique can not be performed on the leg that has had a total knee replacement, but if the other leg meets the inclusion criteria the subject can perform the study on the non- reconstructed leg.
* Patients diagnosed with malignancy over the stimulating electrode site (thigh and knee).
* Patients with serious infection near the stimulating electrode sites (thigh and knee)
* Patients have not had a knee injection in the past 2 weeks.
* Patients who are unable to walk a series of 30 meters without a walking assistance device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Quadriceps central activation ratio | 2 and 4 weeks
Quadriceps torque production | 2 and 4 weeks

SECONDARY OUTCOMES:
WOMAC score | 2 and 4 weeks
Visual analog pain score | 2 and 4 weeks
Knee joint kinetics and kinematics | 2 and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ingersoll, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States